CLINICAL TRIAL: NCT01855373
Title: A Randomized, Double-blind, Placebo-controlled Study Comparing the Healthy Levels of Blood Sugar and Endothelial Function of PEAK ATP® With GlycoCarn®, PEAK ATP® and GlycoCarn® Supplementation Versus Placebo
Brief Title: Comparing Blood Sugar Levels and Endothelial Function of PEAK ATP® With GlycoCarn®, PEAK ATP® and GlycoCarn® Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supplement Formulators, Inc. (Industry)
Collaborators: Sigma Tau HealthScience LLC (Unknown); TSI Health Sciences, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CL049
Record Dates: First submitted 2013-05-13; First posted 2013-05-16 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Blood Sugar; Endothelial Function
Keywords: Blood Sugar; Endothelial Function; Blood Vessel Health

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Other): No active ingredient
  Interventions: Other: Placebo
- PEAK ATP® with GlycoCarn® (Active Comparator): Adenosine 5'-Triphosphate Disodium Salt (100mg/capsule)and Glycine Propionyl-L-Carnitine Hydrochloride, USP (500mg/capsule)
  Interventions: Dietary Supplement: PEAK ATP® with GlycoCarn®
- PEAK ATP® (Active Comparator): Adenosine 5'-Triphosphate Disodium Salt (100mg/capsule)
  Interventions: Dietary Supplement: PEAK ATP®
- GlycoCarn® (Active Comparator): Glycine Propionyl-L-Carnitine Hydrochloride, USP (500mg/capsule)
  Interventions: Dietary Supplement: GlycoCarn®

INTERVENTIONS:
Dietary Supplement: PEAK ATP® with GlycoCarn® — PEAK ATP® with GlycoCarn® {Glycine Propionyl-L-Carnitine Hydrochloride, USP (500mg/capsule) and Adenosine 5'-Triphosphate Disodium Salt (100mg/capsule)}: 2 capsules twice daily on an empty stomach
  Arms: PEAK ATP® with GlycoCarn®
Dietary Supplement: PEAK ATP® — PEAK ATP® (Adenosine 5'-Triphosphate Disodium Salt (100mg/capsule): 2 capsules twice daily on an empty stomach
  Arms: PEAK ATP®
Dietary Supplement: GlycoCarn® — GlycoCarn® (Glycine Propionyl-L-Carnitine Hydrochloride, USP (500mg/capsule): 2 capsules twice daily on an empty stomach
  Arms: GlycoCarn®
Other: Placebo — Placebo: 2 capsules twice daily on an empty stomach
  Arms: Placebo

SUMMARY:
To purpose of this study is to assess the effectiveness, safety and tolerability of PEAK ATP® with GlycoCarn®, PEAK ATP® and GlycoCarn® on levels of blood sugar and endothelial function improvement which may lead to improved vascular health.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, parallel design to evaluate the effectiveness, safety and tolerability of the study substances utilized to support improved healthy levels of blood sugar and endothelial function. Each subject will be randomized to receive a specific dose of PEAK ATP® (Adenosine 5'-Triphosphate Disodium Salt)with GlycoCarn® (Glycine Propionyl-L-Carnitine Hydrochloride, USP (United States Pharmacopeia) , PEAK ATP® (Adenosine 5'-Triphosphate Disodium Salt) and GlycoCarn® (Glycine Propionyl-L-Carnitine Hydrochloride, USP )or Placebo twice daily.

Participants will undergo assessment of blood tests, brachial ultrasound for determining the change in flow mediated dilation, body weight, % body fat, BMI, waist/hip circumference and blood pressure.

The primary objective of the study is to evaluate the safety, tolerability and effectiveness of PEAK ATP® with GlycoCarn®, PEAK ATP® and GlycoCarn® on improving levels of blood sugar via assessment of plasma glucose.

Secondary objectives:

1. To assess flow-mediated dilation as determined by brachial ultrasound evaluation.
2. To assess the effect on changes in blood levels of HbA1C, high-sensitivity C-Reactive Protein (hs-CRP), Insulin, Nitric Oxide (NOx), Malondialdehyde (MAL), Soluble Inter-cellular Adhesion Molecule-1 (sICAM-1) and E-Selectin.
3. To assess the effect on body weight, Body Mass Index (BMI), % body fat as measured by skin caliper, waist and hip circumference, and blood pressure.
4. To assess the effect on general and sexual health for males and females as determined through questionnaires.

ELIGIBILITY:
Primary Inclusion Criteria:

* Ambulatory
* Having the following two criteria:

  1. Confirmed as being overweight (BMI of 25.0-39.9)
  2. Confirmed by a baseline fasting blood sugar level between 95.0-125.0 mg/dl with the glucose meter via finger stick OR laboratory evaluation of glucose level between 95.0-125.0 mg/dl
* Having no difficulty with digestion or absorption of food

Primary Exclusion Criteria:

* Having ever received a clinical diagnosis of cardiovascular disease (excluding hypertension), cancer (excluding basal or squamous cell skin cancer), autoimmune disease (such as systemic lupus, rheumatoid arthritis, multiple sclerosis, psoriasis, etc.), gout, seizures, liver or kidney disease, gallbladder disease, thyroid disease, bi-polar disorder, manic depression, schizophrenia, apathetic (inherited) depression, or any other diagnosis that would preclude study participation in the judgment of the investigator/sub-investigator.
* Having ever received a diagnosis of diabetes mellitus, glucose intolerance, or currently taking any medications for either of the aforementioned conditions.
* Having ever had a re-vascularization procedure (bypass, angioplasty or stent placement) or having received an organ transplant, pacemaker, or internal medical device.
* Currently receiving hormone replacement therapy or taking phosphodiesterase type-5 (PDE-5) inhibitors such as Sildenafil, Vardenafil and Tadalafil.
* If taking aspirin, ibuprofen, naproxen or other anti-inflammatory medication(s), cholesterol medications (including statins), an oral contraceptive, blood pressure medications or medications to treat congestive heart failure (including ACE inhibitors, ACE antagonists or diuretics), must have been on a stable dose for greater than 3 months prior to baseline and be willing to remain on stable dose for duration of study.
* If taking any other cardiovascular drugs including but not limited to antiarrhythmics (excluding beta blockers), inotropic agents, antianginals, or digitalis.
* Having had a history of any medical or surgical procedure that would preclude participation in the study in the judgment of the investigator/sub- investigator.
* Having any blood coagulation disorder or vitamin K deficiency.
* History of allergy to any nutritional supplements, herbal remedies, foods, or any of the components in the study products.
* Have no clinically significant abnormalities on the basis of medical history, physical examination, laboratory evaluation and vital signs in the judgment of the investigator and/or sub-investigator.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Mean change in plasma glucose | 90 days

SECONDARY OUTCOMES:
Mean change in flow-mediated dilation | 90 day
Mean change in HbA1C | 90 days
Mean change in high-sensitivity C-Reactive Protein (hs-CRP) | 90 days
Mean change in insulin level | 90 days
Mean change in Malondialdehyde level | 90 day
Mean change in soluble Intercellular Adhesion Molecule-1 (sICAM-1) | 90 days
Mean change in E-Selectin blood level | 90 days
Mean change in body weight | 90 days
Mean change in Body Mass Index (BMI) | 90 days
Mean change in percent body fat | 90 days
Mean change in waist and hip circumference | 90 days
Mean change in blood pressure | 90 days
Assess the safety and tolerability as measured by various laboratory markers, vital signs and adverse events | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven Joyal, M.D., Principal Investigator — Life Extension
Locations (1):
- Life Extension Clinical Research Inc., Fort Lauderdale, Florida, United States

REFERENCES:
- [Background] Abbracchio MP, Burnstock G, Verkhratsky A, Zimmermann H. Purinergic signalling in the nervous system: an overview. Trends Neurosci. 2009 Jan;32(1):19-29. doi: 10.1016/j.tins.2008.10.001. Epub 2008 Nov 12. PMID 19008000
- [Background] Bannwarth B, Allaert FA, Avouac B, Rossignol M, Rozenberg S, Valat JP. A randomized, double-blind, placebo controlled triphosphate in study of oral adenosine subacute low back pain. J Rheumatol. 2005 Jun;32(6):1114-7. PMID 15940776
- [Background] Bloomer RJ, Smith WA, Fisher-Wellman KH. Glycine propionyl-L-carnitine increases plasma nitrate/nitrite in resistance trained men. J Int Soc Sports Nutr. 2007 Dec 3;4:22. doi: 10.1186/1550-2783-4-22. PMID 18053183
- [Background] Bloomer RJ, Tschume LC, Smith WA. Glycine propionyl-L-carnitine modulates lipid peroxidation and nitric oxide in human subjects. Int J Vitam Nutr Res. 2009 May;79(3):131-41. doi: 10.1024/0300-9831.79.3.131. PMID 20209464
- [Background] Coolen EJ, Arts IC, Bekers O, Vervaet C, Bast A, Dagnelie PC. Oral bioavailability of ATP after prolonged administration. Br J Nutr. 2011 Feb;105(3):357-66. doi: 10.1017/S0007114510003570. Epub 2010 Dec 6. PMID 21129239
- [Background] Cortez-Pinto H, Chatham J, Chacko VP, Arnold C, Rashid A, Diehl AM. Alterations in liver ATP homeostasis in human nonalcoholic steatohepatitis: a pilot study. JAMA. 1999 Nov 3;282(17):1659-64. doi: 10.1001/jama.282.17.1659. PMID 10553793
- [Background] Di Carlo, S. E. and Collins, H. L. (June 1, 2001). Submitting illuminations for review. Advan. Physiol.Edu. 25 (2):70-1. http://advan.physiology.org/ cgi/content/full/25/2/70.
- [Background] Evans AM, Fornasini G. Pharmacokinetics of L-carnitine. Clin Pharmacokinet. 2003;42(11):941-67. doi: 10.2165/00003088-200342110-00002. PMID 12908852
- [Background] http://www.cdc.gov/healthyweight/assessing/bmi/adult_bmi/index.html.
- [Background] http://naturaldatabase.therapeuticresearch.com/nd/Search.aspx?pt=100&id=803&fs=ND&searchid=27239640&cs=&s=ND
- [Background] http://www.pharmgkb.org/do/serve?objId=PA164743471&objCls=Drug#tabview=tab1.
- [Background] Jacobs PL, Goldstein ER, Blackburn W, Orem I, Hughes JJ. Glycine propionyl-L-carnitine produces enhanced anaerobic work capacity with reduced lactate accumulation in resistance trained males. J Int Soc Sports Nutr. 2009 Apr 2;6:9. doi: 10.1186/1550-2783-6-9. PMID 19341458
- [Background] Jordan AN, Jurca R, Abraham EH, Salikhova A, Mann JK, Morss GM, Church TS, Lucia A, Earnest CP. Effects of oral ATP supplementation on anaerobic power and muscular strength. Med Sci Sports Exerc. 2004 Jun;36(6):983-90. doi: 10.1249/01.mss.0000128198.97260.8b. PMID 15179168
- [Background] Knowles JR. Enzyme-catalyzed phosphoryl transfer reactions. Annu Rev Biochem. 1980;49:877-919. doi: 10.1146/annurev.bi.49.070180.004305. No abstract available. PMID 6250450
- [Background] Mace, A.E. (1964), Sample Size Determination, New York: Reinhold Publishing Corporation.
- [Background] Tornroth-Horsefield S, Neutze R. Opening and closing the metabolite gate. Proc Natl Acad Sci U S A. 2008 Dec 16;105(50):19565-6. doi: 10.1073/pnas.0810654106. Epub 2008 Dec 10. No abstract available. PMID 19073922